CLINICAL TRIAL: NCT01347437
Title: Improving Antiretroviral Medication Adherence Among HIV-infected Youth: Phase II
Brief Title: Improving Antiretroviral Medication Adherence Among HIV-infected Youth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fenway Community Health (Other)
Collaborators: Boston Children's Hospital (Other); Massachusetts General Hospital (Other); Harvard Medical School (HMS and HSDM) (Other)
Responsible Party: Principal Investigator, Matthew Mimiaga, Research Scientist, Fenway Community Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CFAR Adherence HIV Youth:2
Record Dates: First submitted 2011-04-04; First posted 2011-05-04 (Estimated); Last update posted 2017-04-17 (Actual); Status verified 2017-04

CONDITIONS: HIV Infection
Keywords: HIV; antiretroviral medication; adherence; adolescent
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Condition (No Intervention): In the comparison condition, participants will receive MEMS only.
- Positive STEPS (Experimental): * Participants will receive one on one Positive STEPS counseling sessions (~1 hour sessions per week for 5 weeks).
  * Participants will receive motivational reminders to take medications sent via text message to their cell phones.
  * Participants will receive the Medication Event Monitoring Systems (MEMS) pill cap monitoring device to measure antiretroviral medication adherence.
  Interventions: Behavioral: Positive STEPS

INTERVENTIONS:
Behavioral: Positive STEPS — This intervention is given to patients in the experimental condition only. The Positive STEPS intervention-developed by our team-is based on general principles of cognitive-behavioral therapy as well as more specific principles of motivational interviewing32,33 and problem solving therapy. Informational, problem solving, and cognitive-behavioral STEPS are targeted over 5, in-person, intervention sessions with a PhD-level counselor. The intervention will also include a series of short videos related to the topics that the Positive STEPS intervention covers with participants. Participants in the experimental condition can also choose to receive text messages sent to their cell phone to remind them to take their medication.
  Arms: Positive STEPS

SUMMARY:
HIV is increasing among adolescents and young adults in the US. Antiretroviral medications, when taken correctly (≥ 90% of prescribed doses taken), can vastly improve life expectancy. However, adherence among HIV-infected young people is suboptimal, and few interventions are available to help adolescents adhere to treatment.

The study is a randomized controlled trial (RCT) pilot trial of Positive STEPS (the adapted form of the Life-Steps behavioral intervention) to improve medication adherence among HIV-infected youth. The study will allow us to demonstrate participant acceptance, ability to recruit, feasibility of intervention delivery with study counselors and all study procedures, and initial clinically significant improvement in medication adherence via MEMS caps. This research will lay the groundwork for a federal grant application for a multi-site randomized controlled intervention trial.

DETAILED DESCRIPTION:
Aims:

1. To conduct a randomized controlled pilot test of a behavioral adherence intervention to improve medication adherence among HIV-infected youth aged 13-24. Feasibility of all study procedures and participant acceptability will be assessed.
2. To explore whether the intervention leads to improved medication adherence among youth who receive the intervention, compared to a control group of youth who do not.

40 HIV-infected adolescents will be recruited for a RCT pilot of the Positive STEPS intervention at Fenway Health and Children's Hospital Boston. Participants will be randomized into one of two arms (half and half). Randomization for all participants will occur after the beginning of the week 2 study visit. The duration of the study is 3 months

Randomization:

The investigators will conduct block randomization based on two categories of electronic adherence: 85% or above versus < 85%. All participants will have exhibited some non-adherence in order to be eligible for the study, although they may vary in the extent of non-adherence. Because insufficient information is known about the range of non-adherence in the population to determine the most valid non-adherence cut-off points, the investigators may need to reconsider adherence categories over the course of the pilot study. The investigators will regularly examine the data to determine whether finer adherence categories are needed, and the investigators will adjust the categories if such a determination is made.

Intervention arm:

* Participants will receive one on one Positive STEPS counseling sessions (~1 hour sessions per week for 5 weeks).
* Participants will receive motivational reminders to take medications sent via text message to their cell phones
* Participants will receive the Medication Event Monitoring Systems (MEMS) pill cap monitoring device to measure antiretroviral medication adherence.

Comparison condition arm:

• Participants will receive the Medication Event Monitoring Systems (MEMS) pill cap monitoring device to measure antiretroviral medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* Age 13 to 24 years
* HIV-infected
* Currently taking antiretroviral therapy or prescribed medication for HIV
* Self-reported difficulties adhering to HIV medications in the past 3 months (i.e., <95% compliant)
* If 18-24: Willing and able to provide informed consent
* If 13-17: Parent/guardian willing and able to provide parental permission and participant willing and able to provide assent
* Willing to attend all study visits

Exclusion Criteria:

* If 18-24:Unwilling or unable to provide informed consent
* If 13-17: Parent/guardian unwilling or unable to provide parental permission and participant willing and able to provide assent
* Has severe mental illness requiring immediate treatment (e.g. active psychotic episode) or a mental illness that would limit your ability to participate (e.g. dementia)
* Has severe cognitive limitation that would limit your ability to comprehend the informed consent or assent (see Decisional Capacity Determination SOP)
* Unwilling to attend all study visits

Ages: 13 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 17 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2013-01 (Actual); Study Completion 2013-03-06 (Actual)

PRIMARY OUTCOMES:
Electronically monitored (MEMS) antiretroviral medication adherence | 3 months
  The primary outcome will be antiretroviral medication adherence. Adherence will be measured through the medication event monitoring device(MEMS).

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Mimiaga, ScD, MPH, Principal Investigator — Massachusetts General Hospital and Fenway Health
Locations (3):
- United States (3):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Children's Hospital Boston, Boston, Massachusetts
  - The Fenway Institute, Fenway Health, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No